CLINICAL TRIAL: NCT04244903
Title: Prevalence of Maxillary Labial Frenal Attachments Types and Midline Diastema in Egyptian Children With Fully Erupted Maxillary Permanent Canines
Brief Title: Prevalence of MLFA Types and MD in Egyptian Children With Erupted Canines
Acronym: diastema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Ahmed Saad, Principal Investigator, Cairo University
Other Study IDs: CEBD-CU-2019-12-05
Record Dates: First submitted 2020-01-25; First posted 2020-01-28 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Destructive Attachment of Labial Frenum
Keywords: Midline diastema, Prevalence, Maxillary frenal types

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Descriptive observational cross sectional study Outpatient at faculty of dentistry Cairo university pediatric dentistry department clinic with midline diastema and fully erupted canines will be examined and assess type of frenal attachment to see if correlation present or not

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy children
* Egyptian children with fully erupted canines
* Patient presented for routine evaluation or treatment

Exclusion Criteria:

* Children who exhibited congenital anomalies or orofacial defects
* Children with previous trauma in frenal area which affect its morphology
* Children have previous surgical intervention in labial frenum or in the maxillary anterior region.
* Children have any syndromes or habits that affect the anterior maxillary region.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will be conducted among Egyptian children with fully erupted canines, who regularly attend the outpatient clinic of pediatric dentistry department, Cairo University.
Sampling Method: Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Midline diastema | 1 year
  measuring diastema in millimeters using calibrated ruler

SECONDARY OUTCOMES:
Frenal attachment types | 1 year
  Direct visual method

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Dentistry Cairo University, Cairo, Giza Governorate
  - Asmaa Ahmed saad, Giza

IPD SHARING:
Plan to Share IPD: Undecided